CLINICAL TRIAL: NCT05109442
Title: A Phase 1/2a Open Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of AFM24 in Combination With Atezolizumab in Patients With Selected Advanced/Metastatic EGFR-expressing Cancers
Brief Title: Study to Assess AFM24 in Combination With Atezolizumab in Selected Advanced/Metastatic EGFR-expressing Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely discontinued due to the financial situation of the sponsor and not for safety or efficacy reasons.
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AFM24-102
Record Dates: First submitted 2021-10-01; First posted 2021-11-05 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — atezolizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation Phase (Experimental): The Escalation phase will determine the MTD/RP2D of AFM24 in combination with atezolizumab. A traditional 3+3 design will be used to determine the RP2D.
  Interventions: Drug: AFM24; Drug: Atezolizumab 840 MG in 14 ML Injection
- Expansion Phase (Experimental): The expansion phase will collect preliminary evidence of efficacy and further confirm the safety of AFM24 in combination with atezolizumab.
  Interventions: Drug: AFM24; Drug: Atezolizumab 840 MG in 14 ML Injection

INTERVENTIONS:
Drug: AFM24 — intravenous infusion
Drug: Atezolizumab 840 MG in 14 ML Injection — intravenous infusion

SUMMARY:
AFM24-102 is a Phase 1/2a open-label, non-randomized, multicenter, dose escalation, and expansion study evaluating AFM24 in combination with atezolizumab in patients with selected EGRF-expressing advanced solid malignancies whose disease has progressed after treatment with previous anticancer therapies.

DETAILED DESCRIPTION:
There will be 2 parts in this study: a dose escalation phase (phase 1) and an expansion phase (phase 2a). Patients will qualify to receive the investigational drugs (AFM24 + atezolizumab) in the dose escalation phase or the expansion phase only if they are deemed eligible following the safety lead-in phase. Seven days before the planned first combination treatment, patients will receive a single dose of AFM24 and will be observed for any adverse events for 1 week.

The aim of the dose escalation phase is to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of AFM24 in combination with atezolizumab.

The dose escalation phase will be followed by the expansion phase once the MTD/RP2D of AFM24 in combination with atezolizumab has been determined. The expansion phase of the study is intended to collect preliminary evidence of efficacy and to further confirm the safety of AFM24 in combination with atezolizumab.

The tumor types planned to be studied in the AFM24/atezolizumab combination study will be:

* Non-small cell lung cancer (EGFR-WT), with disease progression after chemotherapy and PD1/PD-L1 targeted therapy
* Gastric/GEJ cancer if intolerant to or with disease progression after standard platinum-based chemotherapy
* Pancreatic/hepatocellular/biliary tract cancer with disease progression after standard of care (SOC) therapy or if there is no appropriate SOC available for their condition
* Advanced or metastatic NSCLC harboring a targetable EGFR kinase domain mutation with disease progression on or after received ≥1 prior lines of treatment for advanced disease, including a Tyrosine-Kinase Inhibitor (TKI) for EGFR mutations

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic EGFR-positive selected cancer types (except for NSCLC)
* Advanced or metastatic NSCLC, EGFR WT: disease has progressed after ≥ 1 prior lines of therapy which must have included a platinum-based doublet in combination with PD1/PD-L1 antibody or must have received an anti-PD1/PD-L1 antibody prior to or after a platinum-based doublet
* Advanced, unresectable, or metastatic gastric/GEJ adenocarinoma: after ≥ 1 prior chemotherapy regimen including a platinum and fluoropyrimidine doublet
* Advanced or metastatic HCC (BCLC C or B not amenable or refractory to locoregional therapy), hepatobiliary-, or pancreatic adenocarcinoma: after ≥1 prior line of an approved SOC therapy for the respective disease type or to whom the available SOC is not appropriate in the opinion of the investigator
* Advanced or metastatic NSCLC harboring a targetable EGFR kinase domain mutation and whose disease has progressed on or after having received ≥ prior TKI approved for EGFR mutated NSCLC. Subjects treated with a 1st or 2nd generation TKI in 1st line who developed a documented T790M mutation must have received a TKI targeting this mutation such as Osimertinib or Lazertinib to be eligible. Subjects must have documentation of EGFR mutated NSCLC as assessed by an approved test using genomic sequencing of tumor or circulation free tumor DNA. The patients should have received a 2nd line of treatment if approved and available or may be enrolled in the study if in the opinion of the investigator it is in the patient's best interest,or the SOC is not appropriate.
* Adequate organ function
* Phase 1: Evaluable or measurable disease per RECIST v1.1
* Phase 2a: Measurable disease per RECIST v1.1

Exclusion Criteria:

* Treatment with systemic anticancer therapy including investigational agent within 4 weeks of the first dose of study drug, 6 weeks for mitomycin C or nitrosoureas, 2 weeks (or 5 half-lives whichever is longer) for using fluorouracil or small molecule targeted drugs, 2 weeks for using traditional Chinese medicine with anti-tumor indication.
* Radiation therapy within 2 weeks before 1st dose of study drug or unresolved toxicity from previous radiotherapy
* History of any other malignancy known to be active, with the exception of completely removed in situ cervical intra-epithelial neoplasia, non-melanoma skin cancer, DCIS, early stage prostate cancer that has been adequately treated, and other cancers from which the patient has been disease free for 3 years or longer
* Currently active in any other clinical study, or administration of other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Morales-Espinosa, MD, Study Director — Affimed GmbH
Locations (16):
- United States (3):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
- Poland (5):
  - Independent Public Teaching Hospital #4 in Lublin, Department of Clinical Oncology and Chemotherapy, Lublin
  - European Health Center Otwock Fryderyk Chopin Hospital, Department of Clinical Oncology, Otwock
  - MED-Polonia, Sp. z o.o. (LLC), Poznan
  - Janusz Korczak Provincial Specialist Hospital in Slupsk Limited Liability Company, Słupsk
  - Maria Sklodowska-Curie - National Research Institute of Oncology, Early Phase Research Department, Warsaw
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (4):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - University Hospital Quiron Madrid, Madrid
  - University Clinic of Navarra - Pamplona, Pamplona
  - Hospital Clinic Universitario Biomedical Research institute INCLIVA, Valencia
- Royal Marsden NHS Foundation Trust - ICR, Sutton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg: Patients aged 18 years or older with documented histologically or cytologically confirmed select advanced or metastatic epidermal growth factor receptor (EGFR)-positive cancers.
  The patients received AFM24 160 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
- Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg: Patients aged 18 years or older with documented histologically or cytologically confirmed select advanced or metastatic epidermal growth factor receptor (EGFR)-positive cancers.
  The patients received AFM24 480 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
- Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg: Patients aged 18 years or older with advanced or metastatic, EGFR-WT expressing NSCLC whose disease has progressed after having received ≥1 prior lines of therapy for advanced disease. Patients must have received at least a platinum-based doublet in combination with an anti--programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PD-L1) antibody or must have received an anti-PD1/PD-L1 antibody prior to or after a platinum-based doublet. Patients with a known actionable driver mutation (other than EGFR mutation) must have received an approved targeted treatment for the respective mutation. The patients should also have received a second line of treatment if approved and available, or they may be enrolled in the study if in the opinion of the Investigator it is in the patient's best interest, or the standard of care (SOC) is not appropriate.
  The patients received AFM24 480 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
- Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg: Patients aged 18 years or older with locally advanced, unresectable, or metastatic gastric or GEJ adenocarcinoma refractory to or, intolerant of, standard therapy. Patients must have received ≥1 prior chemotherapy regimen including a platinum and fluoropyrimidine doublet. The patients should also have received a second line of treatment if approved and available, or they may be enrolled in the study if in the opinion of the Investigator it is in the patient's best interest, or the SOC is not appropriate.
  The patients received AFM24 480 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
- Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg: Patients aged 18 years or older with advanced or metastatic hepatocellular carcinoma (other than fibrolamellar and sarcomatoid subtype; Barcelona Clinic Liver Cancer Stage C disease or Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy), hepatobiliary-, or pancreatic adenocarcinoma. Patients must have been treated with at least 1 previous line of an approved, SOC therapy for the respective disease type or, in the opinion of the Investigator, available SOC is not appropriate. The patients should also have received a second line of treatment if approved and available, or they may be enrolled in the study if in the opinion of the Investigator it is in the patient's best interest, or the SOC is not appropriate.
  The patients received AFM24 480 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
- Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg: Patients aged 18 years or older with advanced or metastatic NSCLC harboring a targetable EGFR kinase domain mutation and whose disease has progressed on or after having received ≥1 prior lines of therapy for advanced disease including ≥1 prior tyrosine kinase inhibitor (TKI) approved for EGFR mutated NSCLC, such as gefitinib, erlotinib, afatinib, dacomitinib or osimertinib. Patients who were treated with a 1st or 2nd generation TKI in 1st line and developed a documented T790M mutation must have received a TKI targeting this mutation such as osimertinib or lazertinib to be eligible. Patients must have documentation of EGFR mutated NSCLC as assessed by an approved test using genomic sequencing of tumor or circulating free tumor DNA. The patients should also have received a second line of treatment if approved and available, or they may be enrolled in the study if in the opinion of the Investigator it is in the patient's best interest, or the SOC is not appropriate.
  The patients received AFM24 480 mg i.v. qw + atezolizumab 840 mg i.v. q2w in 28-day cycles. AFM24 on Day 1, Day 8, Day 15, and Day 22 (a dose could be given as split day dosing over two days) + atezolizumab on Day 1 and Day 15.
Period: Overall Study
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Started | 4 | 6 | 49 | 12 | 11 | 30
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 6 | 49 | 12 | 11 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 5 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 4 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 2
Not completed — Other than listed | 0 | 0 | 9 | 2 | 0 | 8
Not completed — Lack of Efficacy | 3 | 5 | 29 | 10 | 11 | 17

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Total
Number analyzed (Participants) | 4 | 6 | 49 | 12 | 11 | 30 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.3) | 55.0 (20.2) | 64.9 (9.1) | 59.2 (7.5) | 58.3 (12.1) | 64.2 (9.5) | 62.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 13 | 3 | 7 | 20 | 51
  Male | 0 | 2 | 36 | 9 | 4 | 10 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 45 | 12 | 10 | 30 | 107
  Unknown or Not Reported | 0 | 0 | 4 | 0 | 1 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 18 | 0 | 1 | 18 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 4 | 6 | 30 | 12 | 9 | 12 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 0 | 18 | 0 | 0 | 17 | 35
  United States | 0 | 1 | 1 | 0 | 1 | 2 | 5
  Poland | 0 | 0 | 16 | 0 | 3 | 4 | 23
  United Kingdom | 0 | 1 | 4 | 1 | 0 | 1 | 7
  Spain | 4 | 4 | 10 | 11 | 7 | 6 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Incidence of Dose Limiting Toxicities (DLTs) During Cycle 1
Description: The number of patients with dose limiting toxicities (DLTs) in the first cycle, as assessed by the National Cancer Institute Common Technology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: During cycle 1 (each cycle has 28 days)
Population: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 4 | 6
Participants | 0 | 1

2. Primary Outcome: Phase 2a: Overall Response Rate (Complete Response [CR] or Partial Response [PR])
Description: Tumor assessment by RECIST v1.1 by investigator. Best overall response was used to define the Overall Response Rate (CR or PR). Best overall response is CR or PR if a CR or PR assessed at least 42 days after Cycle 1 Day 1 was confirmed by subsequent tumor assessment at least 4 weeks later.
Time Frame: Tumor assessments were conducted during last week of cycle 2, 4, 6, 8, 10, 12 and every 3 cycles thereafter (each cycle has 28 days), up to approximately 97 weeks.
Population: Full Analysis Set (FAS): All patients who completed the Safety Lead-in phase and received any amount of any component of the combination treatments AFM24 and atezolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 43 | 12 | 11 | 28
Participants | 8 | 1 | 1 | 4

3. Secondary Outcome: Incidence of Patients With TEAEs
Description: Number of patients with treatment-emergent adverse events (TEAEs) non-serious or serious
Time Frame: From first drug administration up to 30 (non-serious TEAEs) or 56 (serious TEAEs) days after last dose AFM24, until start of a subsequent anticancer treatment, or data cut-off date, whichever is sooner. Up to approx. 35 (phase 1) and 105 weeks (phase 2a).
Population: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 4 | 6 | 49 | 12 | 11 | 30
Participants | 4 | 6 | 49 | 11 | 11 | 30

4. Secondary Outcome: Incidence of Patients With SAEs
Description: Number of patients with treatment-emergent serious adverse events (serious TEAEs)
Time Frame: From first drug administration up to 56 days after the last dose of AFM24, until the start of a subsequent anticancer treatment, or data cut-off date, whichever is sooner. Up to approximately 35 (phase 1) and 105 weeks (phase 2a).
Population: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 4 | 6 | 49 | 12 | 11 | 30
Participants | 2 | 3 | 30 | 6 | 7 | 15

5. Secondary Outcome: Pharmacokinetics (PK) of AFM24
Description: Maximum plasma concentration (Cmax) on Cycle 1 Day 22
Time Frame: During cycle 1 (each cycle has 28 days)
Population: All subjects who received at least one adequately documented dose of study drug and had sufficient PK measurements at Cycle 1 Day 22 analysed in central lab.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 4 | 35 | 11 | 8 | 20
ng/mL | 73700 (25400) | 269000 (61400) | 207000 (78100) | 207000 (73400) | 175000 (77200) | 250000 (106000)

6. Secondary Outcome: Pharmacokinetics (PK) of AFM24
Description: Minimum plasma concentration (Cmin) Corresponding to Ctrough levels at the end of the dosing interval at Cycle 1 Day 22
Time Frame: During cycle 1 (each cycle has 28 days)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 4 | 36 | 12 | 7 | 19
ng/mL | 16700 (12500) | 105000 (37200) | 56300 (48500) | 73700 (40900) | 71900 (62500) | 93700 (51600)

7. Secondary Outcome: Pharmacokinetics (PK) of AFM24
Description: Area under the concentration-time curve over the dose interval (AUCtau) on Cycle 1 Day 22
Time Frame: During cycle 1 (each cycle has 28 days)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours*microgram /milliLiter
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 3 | 31 | 11 | 7 | 15
hours*microgram /milliLiter | 5760 (919) | 27900 (9780) | 19800 (9660) | 21500 (8620) | 20500 (11400) | 28600 (11900)

8. Secondary Outcome: Pharmacokinetics (PK) of AFM24
Description: Time to Cmax (Tmax) on Cycle 1 Day 22
Time Frame: During cycle 1 (each cycle has 28 days)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 4 | 35 | 11 | 8 | 20
h | 3.15 (0.03) | 3.15 (0.13) | 9.78 (17.9) | 27.9 (24.5) | 8.63 (15.8) | 10.6 (17.4)

9. Secondary Outcome: Frequency of Patients Developing Anti-drug Antibodies (ADAs) Against AFM24
Description: Measurement of ADAs before and during treatment with AFM24 in combination with atezolizumab Patients with at least one ADA-positive result at baseline or post-baseline counted as developing anti-drug antibodies (ADAs) against AFM24
Time Frame: Ph 1 within 2h prior to: each drug intake (Cycle 1), 1st + 3rd drug intake (Cycle 2 onwards) and at EOT, up to 27 weeks. Ph 2a within 2h prior to: 1st drug intake (Cycle 1 and Cycle 3 onwards), 1st + 3rd drug intake (Cycle 2) and at EOT, up to 97 weeks.
Population: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 4 | 6 | 49 | 12 | 11 | 30
Participants | 1 | 2 | 12 | 2 | 3 | 7

10. Secondary Outcome: Phase 1: Overall Response Rate (Complete Response [CR] or Partial Response [PR])
Description: as for outcome 2
Time Frame: Tumor assessments were conducted during last week of cycle 2, 4, 6, 8, 10, 12 and every 3 cycles thereafter (each cycle has 28 days), up to approximately 27 weeks.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 0

11. Secondary Outcome: Phase 2a: Progression-free Survival
Description: Progression-Free Survival (PFS) was defined as (date of first progression - date of first study drug injection)/30.4375. Patients without progression or death were censored. Tumor assessment by RECIST v1.1 by investigator.
Time Frame: From the first treatment received until the first progression disease assessed by investigator or death.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 43 | 12 | 11 | 28
Months | 3.75 [1.91 to 5.85] | 1.94 [1.48 to 8.71] | 1.91 [0.99 to 2.53] | 3.71 [1.87 to 7.46]

12. Secondary Outcome: Phase 2a: Duration of Response
Description: Duration of Response (DOR) was defined as (date of first progression or death - date of first response (unconfirmed))/30.4375. Patients without response were excluded from the analysis. Patients without progression or death were censored. Tumor assessment by RECIST v1.1 by investigator.
Time Frame: From the date of first response (unconfirmed) until progression disease assessed by investigator or death.
Population: All patients from Full Analysis Set (FAS) (=completed the Safety Lead-in phase and received any amount of any component of the combination treatments AFM24 and atezolizumab) who had a response by RECIST v1.1 by investigator assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 8 | 1 | 1 | 4
Months | 9.20 [3.71 to NA] — Not enough events to calculate the data. | NA [NA to NA] — Not enough events to calculate the data. | 3.71 [NA to NA] — Not enough events to calculate the data. | 11.07 [6.54 to NA] — Not enough events to calculate the data.

13. Secondary Outcome: Phase 2a: Clinical Benefit Rate (CR or PR [Any Duration] or Stable Disease Equal or > 24 Weeks)
Description: Tumor assessment by RECIST v1.1 by investigator. Best overall response was used to define the Clinical benefit rate (CR or PR or SD ≥24 weeks). Best overall response is CR or PR if a CR or PR assessed at least 42 days after Cycle 1 Day 1 was confirmed by subsequent tumor assessment at least 4 weeks later. Best overall response is SD if SD or unconfirmed CR or unconfirmed PR at least 42 days after C1D1. Best overall response SD counts for Clinical benefit rate if SD ongoing for at least 24 weeks.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 43 | 12 | 11 | 28
Participants | 11 | 2 | 1 | 8

14. Secondary Outcome: Phase 2a: Disease Control Rate (DCR) (Complete Response [CR] or Partial Response [PR] or Stable Disease [SD])
Description: Tumor assessment by RECIST v1.1 by investigator. Best overall response was used to define the Disease Control Rate (CR or PR or SD). Best overall response is CR or PR if a CR or PR assessed at least 42 days after Cycle 1 Day 1 was confirmed by subsequent tumor assessment at least 4 weeks later. Best overall response is SD if SD or unconfirmed CR or unconfirmed PR at least 42 days after C1D1.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
Number analyzed (Participants) | 43 | 12 | 11 | 28
Participants | 27 | 5 | 2 | 14

ADVERSE EVENTS:
Time Frame: From first drug administration up to 30 (TEAEs) or 56 (SAEs) days after the last dose of AFM24, until the start of a subsequent anticancer treatment, or data cut-off date, whichever is sooner. Up to approximately 35 (phase 1) and 105 weeks (phase 2a).
Description: Safety Analysis Set (SAS): All patients who received at least any amount of AFM24 or atezolizumab.
  Reported in the tables below are the TEAEs (treatment-emergent Adverse Events).
Arm/Group | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg
All-Cause Mortality (participants affected / at risk) | 3/4 | 5/6 | 21/49 | 9/12 | 9/11 | 9/30
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/6 | 30/49 | 6/12 | 7/11 | 15/30
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 48/49 | 11/12 | 11/11 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg (N=4) | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg (N=6) | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg (N=49) | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg (N=12) | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg (N=11) | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg (N=30)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 1 (1) — TEAE
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) — TEAE
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — TEAE
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 2 (2) — TEAE
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — TEAE
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — TEAE
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) — TEAE
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — TEAE
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — TEAE
Hyperthermia malignant (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — TEAE
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) — TEAE
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — TEAE
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — TEAE
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Cohort 1 - AFM24 160 mg + Atezolizumab 840 mg (N=4) | Phase 1 - Cohort 2 - AFM24 480 mg + Atezolizumab 840 mg (N=6) | Phase 2 - Coh. EXP-1 (EGFR-WT NSCLC) - AFM24 480 mg + Atezolizumab 840 mg (N=49) | Phase 2 - Coh. EXP-2 (Gastric or GEJ Adenocarcinoma) - AFM24 480 mg + Atezolizumab 840 mg (N=12) | Phase 2 - Coh. EXP-3 (Hepatocellular,Hepatobiliary,Pancreatic) - AFM24 480 mg + Atezolizumab 840 mg (N=11) | Phase 2 - Coh. EXP-4 (EGFR Kinase Domain Mutation NSCLC) - AFM24 480 mg + Atezolizumab 840 mg (N=30)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 5 (6) | 25 (31) | 9 (11) | 8 (9) | 19 (20) — TEAE
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — TEAE
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Asthenia (General disorders) | 1 (1) | 1 (1) | 7 (9) | 5 (9) | 8 (13) | 5 (6) — TEAE
Fatigue (General disorders) | 0 (0) | 2 (2) | 8 (9) | 1 (1) | 0 (0) | 4 (4) — TEAE
Pyrexia (General disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 2 (3) | 3 (3) — TEAE
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — TEAE
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — TEAE
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — TEAE
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Soft tissue inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 5 (7) | 3 (3) — TEAE
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (3) | 4 (4) — TEAE
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 5 (8) | 1 (1) | 1 (1) | 0 (0) — TEAE
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) — TEAE
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) — TEAE
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1) — TEAE
Ascites (Gastrointestinal disorders) | 3 (8) | 2 (3) | 0 (0) | 2 (4) | 1 (1) | 0 (0) — TEAE
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — TEAE
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Alanine aminotransferase increased (Investigations) | 1 (2) | 3 (5) | 10 (15) | 3 (6) | 0 (0) | 6 (15) — TEAE
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 8 (12) | 3 (6) | 1 (2) | 6 (25) — TEAE
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (13) — TEAE
Amylase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (4) — TEAE
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (6) — TEAE
Lipase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (3) — TEAE
Weight decreased (Investigations) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (2) — TEAE
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — TEAE
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — TEAE
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — TEAE
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — TEAE
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) — TEAE
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Waist circumference increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 4 (7) | 1 (1) | 4 (4) | 3 (3) — TEAE
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (5) — TEAE
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) — TEAE
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (2) — TEAE
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) — TEAE
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) — TEAE
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) — TEAE
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) — TEAE
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (2) — TEAE
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) — TEAE
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4) — TEAE
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) — TEAE
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (2) | 0 (0) — TEAE
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — TEAE
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — TEAE
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — TEAE
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 5 (5) — TEAE
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 3 (3) — TEAE
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) — TEAE
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — TEAE
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 1 (3) | 4 (8) | 1 (16) | 0 (0) | 5 (8) — TEAE
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 3 (3) | 1 (8) | 3 (5) | 2 (2) — TEAE
Lymphopenia (Blood and lymphatic system disorders) | 3 (25) | 2 (3) | 3 (4) | 0 (0) | 2 (4) | 0 (0) — TEAE
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — TEAE
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — TEAE
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — TEAE
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 4 (5) — TEAE
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 1 (10) | 2 (2) — TEAE
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) — TEAE
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — TEAE
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) — TEAE
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 2 (2) — TEAE
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — TEAE
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) — TEAE
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — TEAE
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 4 (11) | 0 (0) | 0 (0) | 2 (2) — TEAE
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 1 (1) | 3 (3) — TEAE
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — TEAE
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — TEAE
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) — TEAE
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) — TEAE
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) — TEAE
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — TEAE
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — TEAE
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) — TEAE
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (4) — TEAE
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — TEAE
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — TEAE
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) — TEAE
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TEAE
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — TEAE

LIMITATIONS AND CAVEATS:
The study was terminated early (early termination submitted to FDA on 12 June 2025). The decision to terminate early was solely based on the company's financial situation and not influenced by safety or efficacy data. The primary completion date, i.e when the criteria for the final analysis according to the protocol are met is: 06 March, 2025. The data snapshot used for the reported results is 07 April, 2025 (not fully cleaned). SDVs performed: 99.7% for Phase 1, 97.1% for Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has the right to review communications for 90 days prior to public release (whereby the sponsor may ask to consider modifications to ensure necessary protection of sponsor's IP). Any publication shall be not made before the first multi-centre publication if the study is a part of a multi-centred clinical trial. Also, if a publication concerns the analyses of data from a multi-centred clinical trial, the communication shall make reference to the relevant multi-centre publication

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT05109442/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05109442/SAP_001.pdf